CLINICAL TRIAL: NCT03253185
Title: An Open Label Study of SC-007 in Subjects With Advanced Cancer
Brief Title: A Study of SC-007 in Subjects With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Benefit/Risk Imbalance
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-310
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer (CRC); Gastric Cancer
Keywords: Cancer; Advanced cancer; Esophagogastric junction (EGJ) cancers; Maximum tolerated dose (MTD); Maximum Tolerated Dose; Pharmacokinetics
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SC-007 (Experimental): SC-007 intravenous (IV) (various doses and dose regimens)
  Interventions: Drug: SC-007

INTERVENTIONS:
Drug: SC-007 — intravenous

SUMMARY:
This is a multicenter, open-label, Phase 1 study in participants with colorectal cancer (CRC) or gastric cancer to study the safety and tolerability of SC-007 and consists of Part A (dose regimen finding) in participants with CRC followed by Part A in participants with gastric cancer. Part B (dose expansion) will enroll participants into separate disease specific cohorts of CRC or gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced metastatic or unresectable advanced colorectal cancer (CRC) or gastric cancer that is relapsed, refractory, or progressive after:
* CRC: at least 2 prior systemic regimens in the metastatic setting, and as appropriate in patients whose tumors are microsatellite instability-high (MSI-H), pembrolizumab as well.
* Gastric cancer (including gastric and EGJ cancers): at least 2 prior systemic regimens in adjuvant, advanced, or metastatic setting and, as appropriate, a human epidermal growth factor receptor 2 (HER2) targeted agent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Any significant medical condition that, in the opinion of the investigator or sponsor, may place the participant at undue risk from the study.
* Has electrocardiogram (ECG) abnormalities that make QT interval corrected (QTc) evaluation difficult.
* Prior exposure to a pyrrolobenzodiazepine or indolinobenzodiazepine based drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | Minimum first cycle of dosing (Up to 21 days)
  DLTs graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Approximately 4 years
  CBR is defined as the proportion of participants with an objective response or stable disease (CR+PR+SD).
Progression Free Survival (PFS) | Approximately 4 years
  PFS time is defined as the time from the participant's first dose of study drug (Day 1) to either the participant's disease progression or death due to any cause.
Observed plasma concentrations at trough (Ctrough) of SC-007 | Approximately 1 year
  Observed plasma concentrations at trough of SC-007
Incidence of Anti-therapeutic Antibodies (ATAs) against SC-007 | Approximately 4 years
  Incidence of ATAs against SC-007
Overall Survival (OS) | Approximately 4 years
  OS is defined as the time from the participant's first dose date to death due to any cause.
Terminal half life (T1/2) of SC-007 | Approximately 1 year
  Terminal half life of SC-007
Objective Response Rate (ORR) | Approximately 4 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of Response (DOR) | Approximately 4 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Time to Cmax (Tmax) of SC-007 | Approximately 1 year
  Time to Cmax of SC-007
Area under the plasma concentration-time curve within a dosing interval (AUC) of SC-007 | Approximately 1 year
  Area under the plasma concentration-time curve within a dosing interval of SC-007
QTcF Change from Baseline | Up to 9 weeks based on 3 cycles of dosing (21-day cycles)
  QT interval measurement corrected by Fridericia's formula (QTcF)
Maximum observed serum concentration (Cmax) of SC-007 | Approximately 1 year
  Maximum observed serum concentration of SC-007

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - Washington University-School of Medicine, St Louis, Missouri
  - Gabrail Cancer Center Research, Canton, Ohio
  - Tennessee Oncology-Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided